CLINICAL TRIAL: NCT01150552
Title: Prospective Studies of Avian Influenza Transmission to Humans in Egypt
Brief Title: Studies of Avian Influenza Transmission to Humans in Egypt
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: EGYFLU XPD09-211; N01AI70005 (NIH)
Record Dates: First submitted 2010-06-22; First posted 2010-06-25 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Avian Influenza
Keywords: Serology; Poultry; H5N1 virus; HPAI virus
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sera will be tested for human antibodies against AI viruses (types H4-H12) using a microneutralization assay. Study sera will be examined for antibodies against human influenza types H1 and H3 using a hemagglutination inhibition procedure.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Poultry exposed individuals: Any individual who had an occupational contact with poultry in the previous five years will be considered exposed. Individuals working on poultry farms, poultry wet markets, or keeping limited numbers of poultry in their backyard, are considered exposed.
- Non-poultry exposed adult controls: Unexposed individuals must have no occupational exposure to poultry in their lifetime and must also not be exposed to poultry purchased from live bird markets.

SUMMARY:
The main focus of the study is:

* To estimate seroprevalence of AI in poultry-exposed and non-exposed human populations.
* To estimate the incidence of AI in poultry-exposed and non-exposed human populations.
* To investigate risk factors associated with AI infections in occupationally-exposed poultry workers.

The secondary objectives of the study:

* To investigate patterns in transmission of AI to household contacts of AI clinical cases
* To isolate AI viruses from acute cases
* To monitor the pathogenicity and disease severity of AI viruses causing human infections

DETAILED DESCRIPTION:
This 4-year prospective cohort study to compare individuals with occupational exposure to poultry with non-poultry exposed adult controls for evidence of incident and previous infections with AI viruses. At the start of this study, study staff will obtain informed consent, and a blood sample will be obtained from study volunteers to establish baseline levels of antibodies against avian influenza types H4-H12. Subjects will be interviewed regarding their exposures, medical history, and behaviors using a close-ended questionnaire specifically tailored for this study. After one year, study subjects will be interviewed again to note any changes in exposure variables. At this time, another blood sample will be obtained and tested for any changes in antibodies' levels. The same procedures will be repeated at the final visit after another year. Exposed individuals will be selected from rural areas where poultry is commonly raised. Non-exposed controls will be selected from urban neighborhoods in Cairo.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to participate by signing a consent/assent form, completing the study questionnaire, and permitting the withdrawal of blood.
* Does not buy poultry from live bird markets (for controls only).

Exclusion Criteria:

* Any known immunosuppressive condition or immune deficiency disease (including HIV infection), or ongoing receipt of any immunosuppressive therapy.
* Any individual with unknown poultry exposure status, or who was exposed to poultry more than 5 years ago.
* Children who are less than 2 years old when baseline enrollment is performed.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Exposed subjects will be enrolled at the rural areas of Egypt where poultry production is located. Controls will be enrolled in urban Cairo. Households will be selected from neighborhoods without live bird markets close to the location of the NRC. All members of a household will be enrolled. Cohort of exposed subjects will be assembled from villages from 3 governorates in this area as well as 2 governorates south of Cairo where human cases of AI were reported. Hence, 5 villages will make up 5 field sites. From each village, the team will enroll 150 individuals with exposure to poultry. The control group, i.e., individuals not occupationally exposed to poultry, will be enrolled from urban Cairo, the capital of Egypt.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Measure antibodies in sera collected from poultry-exposed and non-exposed individuals | 4 years
  Prevalence rates will be measured by the presence of antibodies against AI viruses of types H4-H12 using a microneutralization assay.
Draw 3 annual serum samples from each individual and record any increase in the antibody titers against AI viruses. | 4 years
  Incidence rates will be assessed based on a 2-fold increase of antibody titers between baseline and follow-up and between follow-up and the final visit.
Risk or protective factors correlated with infection will be measured using the enrollment questionnaire. | 4 years

SECONDARY OUTCOMES:
Obtain nasal and naso-pharyngeal swabs from subjects reporting ILI symptoms and confirm the presence of influenza by a rapid test. | 4 years
  Obtain swabs from the household contacts of individuals with a confirmed influenza A infection and test them for the presence of influenza A viruses
To send RT-PCR positive specimens collected from subjects reporting ILI symptoms to the hospital in order to isolate and characterize the virus. | 4 years
Collect data on disease pathogenicity and severity of symptoms from subjects reporting ILI and obtain a blood sample to isolate and study peripheral blood mononuclear cells. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ghazi Kayali, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- National Research Centre, Giza, Egypt

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols